CLINICAL TRIAL: NCT00322010
Title: A Randomized Trial of Early Physical and Occupational Therapy in Mechanically Ventilated, Critically Ill Patients
Brief Title: Early Directed Physical Therapy in the Management of Mechanically Ventilated Patients in a Medical Intensive Care Unit
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13766B
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Mechanically Ventilated Patients
Keywords: mechanical ventilation; physical therapy; occupational therapy; mobilization; clinical protocols; ICU acquired weakness; critical illness myopathy; muscle atrophy; intensive care unit; randomized controlled trial
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early PT OT (Experimental): Early PT/OT Therapy assessments to begin on the first day that consent is obtained. Therapy is delivered by a team consisting of a physical and occupational therapist and coordinated with daily sedative interruption.
  Interventions: Procedure: early PT OT
- Standard Care (No Intervention): PT/OT delivered as ordered by the primary ICU team

INTERVENTIONS:
Procedure: early PT OT — 1. Passive range of motion exercises for all limbs in patients who remain unresponsive despite sedative interruption (ten repetitions in all cardinal directions).
  2. Sessions began with active assisted and active range of motion exercises in the supine position.
  3. If tolerated, treatment is advanced to bed mobility activities, including transferring to upright sitting.
  4. Sitting balance activities are followed by participation in activities of daily living (ADLs) and exercises that encourage increased independence with functional tasks.
  5. The session progresses to transfer training, and finally pre-gait exercises and ambulation.
  6. Progression of activities is dependent on patient tolerance and stability.
  7. Therapy intervention continues on a daily basis throughout the patient's hospital stay until he/she returns to prior level of function or is discharged.
  Arms: Early PT OT

SUMMARY:
To study all ICU patients with an independent baseline functional status, who experience a critical illness requiring intubation and mechanical ventilation, evaluating the role of protocol-directed, early physical and occupational therapy on the incidence of critical illness associated functional debilitation. Our goal is to hasten the recovery of independent physical functioning as well as to reduce ICU delirium in the group of patients who begin this intervention from the earliest hours of ventilator dependence.

ELIGIBILITY:
Inclusion Criteria

1. Patients intubated and mechanical ventilated for < 72 hours
2. Age > 18 years
3. Baseline independent functional status as assessed by a Barthel Index score > 70 collected from a proxy reflecting baseline health 2 weeks prior to critical illness

Exclusion Criteria

1. Rapidly evolving neurological/neuromuscular disease
2. Cardiac arrest
3. Irreversible conditions with six month mortality estimated at > 50%
4. Elevated intracranial pressure
5. Multiple absent limbs (precluding complete musculoskeletal examination)
6. Enrollment in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2005-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Number of patients returning to independent functional status: defined as ability to perform 6 activities of daily living (ADL's)(bathing, dressing, eating, grooming, transfer from bed to chair, toileting) and independent ambulation | Hospital Discharge

SECONDARY OUTCOMES:
Number of hospital days with delirium | Hospital discharge
Number of days alive and breathing without assistance (ventilator-free days) | during 28-day study period
length of stay | ICU and Hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: John P Kress, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324